Cover page with the Official Title of the study:

Effectiveness of a Self-applied Positive Psychology Online Intervention Program "Mental Health COVID-19" in Mexican population: A Randomized Controlled Trial.

Date: May 15th of 2020



## Informed consent

A group of researchers from the International University of Valencia, the Autonomous University of Ciudad Juárez (UACJ) and the Autonomous University of Mexico (UNAM), we are conducting a study in order to know the current status of the psychosocial and health problems faced with the contingency that the Mexican population is currently suffering due to SARS-CoV-2 (COVID-19) and to implement a brief online intervention based on Positive Psychology. The intervention is made up of 15 interconnected modules to which you will have access when registering on the platform.

To register on the platform, only an email is required, and you do not have to provide sensitive or personally identifiable information such as your name at any time. The results of this research will be analyzed for research purposes and, therefore, can be published in journals, scientific books or disseminated by other means to the scientific community, taking care at all times of the confidentiality and anonymity of the data of the participants. This study has the approval of the ethics committee of ELPAC University of Behavioral Sciences. Approval date May 01, 2020. Identification number: Folio N.2008. It is important to mention that you will not be asked for any sensitive data or your name, in addition to the fact that the intervention will always be completely free.

For this reason, to start we ask you to answer a series of questions that will be presented below, a task that will take you around 30-35 minutes. If there is a question that you do not understand, please report it to us and continue with the next question, the important thing is that you answer what exactly happens in your case, because that is precisely what we want to know. There are no right or wrong questions, so please answer with the utmost sincerity.

## The instruments to answer are:

- 1. Scale collective traumatic events pineda, guerrero, pinilla, estupiñán (2002). Validation and adaptation by chávez-valdez, esparza-del villar and rivers velasco-moreno (2020)
- 2. Diffuse fear scale. (social anxiety) ruiz, j, i. (2002). Adapted by Chávez and Ríos Velasco (2018)
- 4. Collective efficacy scale. Ruiz, j, i. (2002). Adapted by Chávez and Ríos Velasco (2018)
- 5. Self-assessment inventory: state-trait anxiety (IDARE) (Spielberger, Díaz-Guerrero, 1975)
- 6. Scale of suicidal thoughts (Beck, 1979)

- 7. General Anxiety Disorder GAD-7. (Spitzer, Kroenke, Williams, Löwe, 2006)
- 8. Depression scale. (Beck, 1996)
- 9. Pittsburgh sleep quality index. (Buysse, 1989)

If you agree with what is proposed, please click on accept, otherwise you can close your internet window. In this application, you indicate that you agree to voluntarily participate in this research that we are conducting and, therefore, willing/complete the questionnaires.

I accept and commit to respect the following standards in order to provide knowledge, progress, and research on the health of the Mexican population that is being exposed to the contingency due to the COVID-19 pandemic, therefore, I declare that:

- I have been able to ask questions about the study
- •I have received enough information about the study
- I can contact the people who are applying this series of questionnaires to dispel my doubts regarding the research.

I understand that my participation is voluntary and that I can withdraw from the study:

- 1. Anytime
- 2. Without having to explain
- 3. Without this affecting my integrity as a person

I freely agree to participate in the study

## Benefits:

If you accept their participation, you will join a psychosocial and health support network, where you will receive free Psychological counseling through a program of 15 interactive modules and a chat service which will be attended by Psychologists supervised by the researchers of this project and which It is intended to clarify any doubts you may have regarding the contents of the modules or tasks to be performed.

For more questions, you can contact us by mail at admin@saludmentalcovid.com or Dr. Alejandro Domínguez Rodríguez, principal investigator, and coordinator of this project:

alejandro.dominguez.r@campusviu.es

I freely agree to participate in the study: